CLINICAL TRIAL: NCT03930381
Title: Adapting and Expanding the Algorithmic Software Tool to Help Manage Asthma (ASTHMAXcel) for Youth With Asthma
Brief Title: Adapting and Expanding the Asthma-Educator App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-9083
Record Dates: First submitted 2019-04-05; First posted 2019-04-29 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Study will eventually compare health outcomes between a group given the ASTHMAXcel intervention and a group given Usual Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): This group will download the ASTHMAXcel application and use it for the duration of the study
  Interventions: Other: ASTHMAXcel App
- Usual Care Arm (No Intervention): This group will just receive normal provider care

INTERVENTIONS:
Other: ASTHMAXcel App — ASTHMAXcel includes interactive games, educational videos, quizzes and personalized feedback to teach different aspects of asthma management.
  Arms: Intervention Arm

SUMMARY:
This project seeks to test and refine an adapted/expanded version of a previously created ASTHMAXcel app.

DETAILED DESCRIPTION:
The study will test the adapted app on participants ages 15-21 (recruited from outpatient primary and specialty care sites at Montefiore) with asthma, for a period of 4 and a half months, and will conduct formative and summative evaluation of the application's functionality and usability. The investigators will also be collecting process and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking individuals between 15-21
* Persistent asthma (diagnosis made by a healthcare provider)
* On a daily controller medication
* Able to give informed consent
* Smartphone (iOS or Android) access

Exclusion Criteria:

* Use of oral corticosteroids in the 2 weeks prior to the baseline visit
* Pregnancy
* Severe psychiatric or cognitive problems that would prohibit an individual from understanding and completing the protocol
* Patients that previously received the ASTHMA-Educator application

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Asthma Control to 3 Month Asthma Control | Post-Refinement Baseline, 3 Months
  Asthma symptom burden as measured by the Asthma Control Test
  Score Scale: 5 (min = worse); 25 (max = better outcome)
Change from Baseline Asthma Control to 3 Month Asthma Control | Post-Refinement Baseline, 4 Months
  Asthma symptom burden as measured by the Asthma Control Test
  Score Scale: 5 (min = worse); 25 (max = better outcome)

SECONDARY OUTCOMES:
Asthma Symptom Perception | Week 2, Week 4 , Week 6 (Pre and Post Refinement)
  Ability of participants to perceive their asthma symptoms by using the ASTHMAXcel app and a peak flowmeter
Asthma Knowledge | Post-Refinement Baseline, 3 Month
  Will use the Child Asthma Illness Representation Survey (AIRS) to asses patients knowledge on asthma as well as their attitudes towards their condition.
  Score Scale: 4 (min = worse outcome); 20 (max = better outcome)
Medication Adherence | Post-Refinement Baseline, 3 Month
  Self-reported adherence by patient using Medication Adherence Report Scale
  Score Scale: 10 (min = worse outcome); 50 (max = better outcome)
Asthma Quality of Life | Post-Refinement Baseline, 3 Month
  Quality of life of participants, measured by mini-Asthma Quality of Life Questionnaire
  Score Scale: 15 (min = worse outcome); 105 (max = better outcome)
Emergency Department Visits | Post-Refinement Baseline, 3 Month
  Self-Reported Emergency Department (ED) visits
Patient Satisfaction | Post-Refinement Baseline, 3 Month
  Patient satisfaction with study measured by the Client Satisfaction Questionnaire-8
  Score Scale: 8 (min = worse outcome); 32 (max = better outcome)
Patient Interface Satisfaction | Post-Refinement Baseline, 3 Month
  Patient satisfaction with ASTHMAXcel app interface measured by Questionnaire for User Interface Survey (QUIS)
  Score Scale: 0 (min = worse outcome); 261 (max = better outcome)
  Answers scale from 0 (terrible/hard to understand)) to 9 (wonderful/easy to understand)
Patient Usage | Baseline, 3 Month
  Time spent on app and different screens of app, measured using Google Analytics
Health Literacy | Post-Refinement Baseline
  Ability for patients to comprehend Newest Vital Sign screening tool

CONTACTS AND LOCATIONS:
Overall Officials: Sunit Jariwala, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan A, De Simoni A, Wileman V, Holliday L, Newby CJ, Chisari C, Ali S, Zhu N, Padakanti P, Pinprachanan V, Ting V, Griffiths CJ. Digital interventions to improve adherence to maintenance medication in asthma. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD013030. doi: 10.1002/14651858.CD013030.pub2. PMID 35691614